CLINICAL TRIAL: NCT05057351
Title: Randomized, Double Blind, Clinical Study for Evaluating the Efficacy and the Tolerability of a Cosmetic Active Ingredient Intended for Subjects With Atopic Dermatitis. Controlled Study vs Placebo
Brief Title: A Controlled Study to Evaluate the Efficacy and the Tolerability of a Cosmetic Active Ingredient Intended for Subjects With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Greenpharma S.A.S. (Other)
Collaborators: Complife Italia S.r.l (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H.E.HU.AD.NSO05.066.05.00
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Mild to Moderate Atopic Dermatitis

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, placebo-controlled, parallel group study, carried on 2 groups of 22 subjects.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active ingredient (Experimental): Isopentenyltheophylline 0.44% + Glycerin 4.56%
  Interventions: Other: Isopentenyltheophylline 0.44% + Glycerin 4.56%
- Placebo (Placebo Comparator): Glycerin 4.56%
  Interventions: Other: Glycerin 4.56%

INTERVENTIONS:
Other: Isopentenyltheophylline 0.44% + Glycerin 4.56% — Application of topical cream twice a day on the area affected by Atopic Dermatitis
  Arms: Active ingredient
Other: Glycerin 4.56% — Application of topical cream twice a day on the area affected by Atopic Dermatitis
  Arms: Placebo

SUMMARY:
Evaluation of safety and clinical efficacy of an active ingredient versus placebo for the treatment of mild to moderate Atopic Dermatitis (AD) adults.

ELIGIBILITY:
Main Inclusion Criteria:

* Good general health
* Phototype I to IV
* Mild to moderate SCORAD (between 15 and 25)

Main Exclusion Criteria:

* Pregnant/breastfeeding female or who have planned a pregnancy during the study period
* Positive history for atopy or hypersensitive skin
* Subjects under systemically pharmacological treatment
* Subjects under locally pharmacological treatment on the skin area monitored during the test
* Subjects with congenital or acquired immunodeficiency
* Subjects under treatment with food supplements which could interfere with the functionality of the product under study
* Subjects which show other skin alterations on the monitored area except for acne lesions
* Subjects with known or suspected sensitization to one or more test formulation ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in severity of Atopic Dermatitis as assessed using the SCORing Atopic Dermatitis (SCORAD) | 7, 14 and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Roveda, MD, Principal Investigator — Complife Italia S.r.l
Locations (1):
- Complife Italia S.r.l., San Martino Siccomario, Italy

IPD SHARING:
Plan to Share IPD: No